CLINICAL TRIAL: NCT04765839
Title: Community-Engaged Bidirectional Pandemic Crisis and Emergency Risk Communication With Minority Populations
Brief Title: Community-Engaged Bidirectional Pandemic Crisis and Emergency Risk Communication With COVID-19 Vaccine Messages to Minority Populations
Acronym: CERC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark L Wieland, Chair, Community Internal Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-000205
Record Dates: First submitted 2021-02-02; First posted 2021-02-23 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Vaccine Preventable Disease
Keywords: hesitancy
MeSH Terms: conditions — Vaccine-Preventable Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomization outcomes will not be disclosed to participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm - Receives COVID-19 Vaccine messages (Experimental): Group to receive COVID-19 Vaccine messages during the first two weeks of the study.
  Interventions: Other: Educational, culturally appropriate COVID-19 messages
- Delayed Intervention Arm (Experimental): Group to receive COVID-19 Vaccine messages during the last two weeks of the study.
  Interventions: Other: Educational, culturally appropriate COVID-19 messages

INTERVENTIONS:
Other: Educational, culturally appropriate COVID-19 messages — Educational, culturally appropriate COVID-19 messages will be developed and shared by RHCP.

SUMMARY:
A cluster randomized trial will be conducted prior to widespread vaccine availability to the general public. Community-informed COVID-19 vaccine messages will be disseminated to participants. At baseline, 2 weeks and 4 weeks, the study team will survey participants to assess knowledge and attitudes about COVID-19 vaccines, including intention to be vaccinated.

DETAILED DESCRIPTION:
A cluster randomized trial with 80 participants from the social networks of 8 CLs will be conducted prior to widespread vaccine availability to the general public. Four CLs and social networks (cluster of 10 per network) will be randomly assigned to receive the intervention immediately or after a delay of 2 weeks. Intervention participants will be invited to a closed social media group on the platform of their choice. CLs, selected for trustworthiness within vulnerable populations, will disseminate community-informed COVID-19 vaccine messages to members of their social networks and engage in bidirectional communication with CEnR partners to refine messages. At baseline, 2 weeks and 4 weeks, participants will be surveyed to assess knowledge and attitudes about COVID-19 vaccines, including intention to be vaccinated.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification within a CLs social network
* Age 18 or greater
* Functional internet access.

Exclusion Criteria:

* Does not self-identify within a CLs social network
* Is under the age of 18
* Does not have functional internet access.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-04-03 (Actual); Study Completion 2021-04-03 (Actual)

PRIMARY OUTCOMES:
COVID-19 attitudes | 4 weeks
  Related to perceived susceptibility and preventive measures will be assessed through 3 survey instruments, based on 7-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mark, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No